CLINICAL TRIAL: NCT05903287
Title: A Study to Evaluate Accuracy and Validity of Chang Gung Pleural Effusion Detection Software Compared With Reference by Qualified Physicians
Brief Title: Validity of Pleural Effusion Detection Software
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202300606A5
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-06

CONDITIONS: Pleural Effusion
Keywords: artificial intelligence
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Software diagnosis: Software diagnosis with gold standard of 3 specialist physicians' interpretation.
  Interventions: Device: Chang Gung Pleural Effusion Detection Software

INTERVENTIONS:
Device: Chang Gung Pleural Effusion Detection Software — The Chang Gung Pleural Effusion Detection Software is an independent software as a medical device, which inputs digital Chest X-Ray to automatically detect whether there is a pleural effusion. The inferred results output by this software can assist clinicians or professional medical personnel to identify whether a patient has pleural effusion.
  This product is only used to analyze the digitized Chest X-Ray DICOM of patients over 20 years old and under 100 years old.

SUMMARY:
The Chang Gung Pleural Effusion Detection Software is a medical software that can automatically detect whether there is a pleural effusion in Chest X-Ray. The purpose of this study is to verify whether the Chang Gung Pleural Effusion Detection Software can correctly identify patients with pleural effusion in Chest X-Ray. The results of the software analysis will be used for the performance of the software on the primary and secondary outcomes.

DETAILED DESCRIPTION:
This clinical trial is a retrospective study. DICOM images of de-identified Chest X-Ray were collected from 6 hospitals of Chang Gung Memorial Hospital from January 1, 2018 to December 31, 2020. After confirming that the Chest X-Ray that meet the inclusion and exclusion criteria are correct, 282 samples will be sampled for this test, including 141 images with pleural effusion and 141 images without pleural effusion. The image must be in DICOM format.

Then, 3 specialists physicians interpret 282 samples whether there were pleural effusion, and the result was the standard of this study (Reference standard). After determining the reference standard of each Chest X-Ray, the 282 samples were input into the Chang Gung Pleural Effusion Detection Software, and analyzed by the primary and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* The case were over 20 years old and under 100 years old.
* DICOM format.
* Brand model of Canon.
* DICOM resolution length range (700-3400 pixels), width range (490-3600 pixels).
* poster-anterior view(PA-view) of chest X-ray

Exclusion Criteria:

* The chest X-ray contains items that affect interpretation, such as chest tubes, endotracheal tubes, and heart rhythm regulators, but does not include patches and circuits used in electrocardiograms.
* The chest X-ray that are difficult to interpret due to poor image quality.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective study, and the data comes from the Chang Gung Medical Research Database(CGRD) which was an database form 6 hospitals of Chang Gung Memorial hospital. According to inclusion and exclusion criteria, Chest X-ray data from the database during 2018.01.01~2020.12.31 was collected.
Sampling Method: Probability Sample
Enrollment: 282 (Estimated)
Dates: Start 2023-06-17 (Actual); Primary Completion 2023-11-23 (Actual); Study Completion 2024-08-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | baseline
  The rate of test results that correctly indicate the presence.

SECONDARY OUTCOMES:
Specificity | baseline
  The rate of test results that correctly indicate the absence.
Area Under the receiver operating characteristic Curve | baseline
  A graphical plot that illustrates the diagnostic ability of a binary classifier system as its discrimination threshold is varied.

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Fu Kuo, MD/Ph.D, Study Chair — Associate Professor and Director Division of Rheumatology
Locations (1):
- Chang Gung memorial hospital, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahn JS, Ebrahimian S, McDermott S, Lee S, Naccarato L, Di Capua JF, Wu MY, Zhang EW, Muse V, Miller B, Sabzalipour F, Bizzo BC, Dreyer KJ, Kaviani P, Digumarthy SR, Kalra MK. Association of Artificial Intelligence-Aided Chest Radiograph Interpretation With Reader Performance and Efficiency. JAMA Netw Open. 2022 Aug 1;5(8):e2229289. doi: 10.1001/jamanetworkopen.2022.29289. PMID 36044215
- [Background] Lachin JM. Properties of simple randomization in clinical trials. Control Clin Trials. 1988 Dec;9(4):312-26. doi: 10.1016/0197-2456(88)90046-3. PMID 3203523
- [Background] Suresh K. An overview of randomization techniques: An unbiased assessment of outcome in clinical research. J Hum Reprod Sci. 2011 Jan;4(1):8-11. doi: 10.4103/0974-1208.82352. PMID 21772732
- [Background] Lim CY, In J. Randomization in clinical studies. Korean J Anesthesiol. 2019 Jun;72(3):221-232. doi: 10.4097/kja.19049. Epub 2019 Apr 1. PMID 30929415